CLINICAL TRIAL: NCT05970705
Title: A Randomized, Controlled, Multicenter Phase II Trial of Regorafenib Combined With Trifluridine/Tipiracil Versus Regorafenib Monotherapy in Patients With Metastatic Colorectal Cancer Who Failed at Least Two Lines of Systematic Therapy
Brief Title: Regorafenib Combined With TAS-102 Versus Regorafenib Monotherapy in Third or Later Line Therapy of mCRC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Weijian Guo, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDZL-REGOT
Record Dates: First submitted 2023-07-03; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer; regorafenib; TAS-102; Trifluridine/Tipiracil
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib; trifluridine tipiracil drug combination

STUDY DESIGN:
Intervention Model Description: controlled, randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Regorafenib+TAS-102 combination therapy (Experimental): Regorafenib 80mg ,orally, once a day, d1-28, every 28 days, TAS-102，35mg/m2, orally，twice a day, d1-5 & d15-19，every 28 days
  Interventions: Drug: Regorafenib; Drug: Trifluridine/Tipiracil
- B：Regorafenib monotherapy (Active Comparator): Regorafenib, 120mg orally, once a day, d1-21, every 28 days (If the patient's body surface area is less than 1.5m2, the starting dose of regorafenib is 80mg)
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib — this anti-angiogenesis targeting drug is one of the standard third-line treatment options for patients with metastatic colorectal cancer
  Other Names: Stivaga
Drug: Trifluridine/Tipiracil — this chemotherapeutic drug is also one of the standard third-line treatment options for patients with metastatic colorectal cancer
  Other Names: TAS-102
  Arms: A: Regorafenib+TAS-102 combination therapy

SUMMARY:
The purpose of this study is to evaluate the clinical benefit of regorafenib combined with TAS-102 compared with regorafenib monotherapy in patients with metastatic colorectal cancer who have failed at least two lines of treatment, to explore the rationality of this combination therapy strategy and to obtain relevant survival and safety data.

DETAILED DESCRIPTION:
Based on the current diagnostic and treatment guidelines, regorafenib and TAS-102 monotherapy are both standard third-line treatment options for patients with metastatic colorectal cancer (mCRC), yet the overall treatment sequence or preference is not clear. A retrospective study directly compared the efficacy of regorafenib and TAS-102 monotherapy for third-line treatment of mCRC, and found similar efficacy between the two treatments. However, the benefits of current third-line monotherapy for mCRC are still limited. Patients who receive oral regorafenib monotherapy have an ORR of less than 5%, disease control rate of 50-60%, and TAS-102 has an ORR of 1.1%-1.6% and a disease control rate of less than 50% in third-line treatment of mCRC. These drugs have limited prolongation of progression-free survival (PFS), and disease progression and drug resistance often occur shortly after medication use. Most mCRC patients have a high tumor burden during third-line treatment, and how to improve the remission rate of treatment, improve patients' quality of life due to high tumor burden, increase disease control, and further bring better survival benefits is still a big challenge for third-line treatment. Regorafenib and TAS-102 have different mechanisms of action and different adverse reaction spectra. When the two drugs are used in combination, they may complement each other in terms of efficacy and are also less likely to have toxic effects.

In the RECOURSE study, 17% of patients in the TAS-102 treatment group had received prior treatment with regorafenib. Subgroup analysis showed that the efficacy of TAS-102 was not dependent on whether or not the patient had previously received regorafenib treatment. Therefore, the combination of regorafenib and TAS-102 may be a valuable treatment option for refractory mCRC. However, there is little clinical research data on whether the combination therapy could further improve efficacy and prolong patient survival compared to monotherapy. In 2021, a phase Ib small-sample study from Germany explored the combined use of regorafenib and TAS-102 in third-line treatment of mCRC. The study included 12 patients who received combined treatment with regorafenib and TAS-102 in third-line treatment. After a 3+3 dose-exploration trial, three cases of DLT were all grade 3 hypertension related to regorafenib. The combination of TAS-102 25 mg/m2 twice daily and regorafenib 120 mg was well tolerated, with a median PFS of 3.81 months (95% CI: 1.51-5.2), and a median OS of 11.1 months (95% CI: 2.3-18.2). The results of this early-phase clinical trial suggest that compared to regorafenib monotherapy in the CORRECT study with a median PFS of less than two months and a median OS of less than seven months, the third-line combination treatment of regorafenib and TAS-102 may potentially provide patients with greater clinical benefits. In conclusion, the combination therapy of regorafenib and TAS-102 may be further explored and studied for late-stage colorectal cancer in third-line or after third-line treatment.

The aim of this study is to evaluate the clinical benefits and safety of the combination of regorafenib and TAS-102 compared to regorafenib monotherapy in patients with advanced colorectal cancer who have failed second-line or later treatments. The efficacy and safety of the combination therapy will be fully evaluated, and explorations of efficacy, PFS, OS, safety, and related biomarkers associated with the combined treatment of regorafenib and TAS-102 will be conducted.

ELIGIBILITY:
A total of 101 patients with metastatic colorectal cancer who meet the inclusion criteria and do not meet the exclusion criteria for receiving third-line or later-line therapy will be randomly assigned to receive corresponding treatment in a 1:1 ratio.

Inclusion Criteria:

The subjects must meet all of the following criteria to be eligible for this study:

1. Patients with histologically confirmed recurrent/metastatic colorectal adenocarcinoma.
2. Patients who have failed at least one prior standard first- or second-line therapy, including fluoropyrimidine-based therapy, oxaliplatin, irinotecan, and bevacizumab. Treatment failure is defined as either radiographic evidence of disease progression or unacceptable toxicity during treatment or within three months following completion of therapy.

   (Note: a. each line of therapy should include at least one or more chemotherapy agents administered for at least one cycle; b. adjuvant/neoadjuvant therapy is allowed. If relapse or metastasis occurs during or within six months after completion of adjuvant/neoadjuvant therapy, it is considered a failure of first-line chemotherapy for progressive disease. c. For patients with RAS/RAF wild-type tumors, the use of an EGFR inhibitor is not required.)
3. At least one measurable lesion, with the longest diameter ≥10 mm on spiral CT or ≥20 mm on conventional CT (RECIST 1.1 criteria).
4. ECOG performance status of 0-2.
5. Life expectancy of ≥12 weeks.
6. Adequate bone marrow, hepatic, and renal function measured within the screening period prior to randomization: absolute neutrophil count (ANC) ≥1.5 × 109 /L, hemoglobin ≥ 8.0 g/dL, platelet count ≥ 75 × 109 /L, total bilirubin <1.5 × ULN, ALT and AST <2.5 × ULN (≤5 × ULN for patients with liver involvement), serum creatinine ≤1.5 × ULN, and creatinine clearance ≥50 mL/min.
7. Women of childbearing potential must use effective contraception.
8. Voluntarily participating in this study, signing the informed consent form, understanding the purpose of the study and the necessary procedures, and willing to participate in this study.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study:

1. Proteinuria ≥2+ on dipstick or 24-hour urinary protein ≥1.0 g/24 h.
2. Abnormal coagulation function (PT>16s, APTT>43s, TT>21s, Fbg<2g/L), bleeding tendency, or receiving thrombolysis or anticoagulation therapy.
3. Patients at risk of gastrointestinal bleeding, including those with active digestive ulcers and fecal occult blood (++) and those with histories of black stools or hematemesis within three months.
4. Receiving systemic antitumor therapy, including chemotherapy, signal transduction inhibitors, or immune therapies, within three weeks prior to screening.
5. Patients with uncontrolled hypertension (systolic blood pressure >140 mmHg, diastolic blood pressure >90 mmHg) despite antihypertensive medication, grade I or higher coronary heart disease, grade I or higher arrhythmia (including QTc interval prolongation with ≥450 ms for men and ≥470 ms for women), or grade I or higher heart failure.
6. Patients with a history of thrombotic or embolic events requiring treatment within the preceding six months.
7. Patients who have received radiation therapy targeting the selected target lesion.
8. Symptomatic brain or meningeal metastasis.
9. Uncontrolled pleural or peritoneal effusion.
10. Receiving kidney dialysis.
11. Serious or uncontrolled infection.
12. Pregnant or lactating women or women of childbearing potential without adequate contraception.
13. Multiple factors affecting oral drug administration (dysphagia, chronic diarrhea, and bowel obstruction).
14. Patients who have been treated with small molecule tyrosine kinase inhibitors containing VEGFR (such as apatinib, fruquintinib, anlotinib, and lenvatinib).
15. Patients who have been treated with TAS-102.
16. Participation in another clinical study within four weeks prior to screening.
17. Patients with comorbidities that could seriously endanger patients' safety or affect their completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-07-04 (Estimated); Study Completion 2026-07-04 (Estimated)

PRIMARY OUTCOMES:
PFS | from the time signing of ICF until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  progression free survival

SECONDARY OUTCOMES:
OS | from the time signing of ICF until the date of death from any cause, assessed up to 36 months
  overall survival
ORR | the rate of patients with CR and PR, through study completion, an average of 1 year
  objective response rate
DCR | the rate of patients with CR, PR and SD, through study completion, an average of 1 year
  disease control rate
DOR | the time between the first tumor evaluation for CR or PR and the first evaluation for PD(Progressive Disease) or death from any cause, assessed up to 36 months
  duration of response

OTHER OUTCOMES:
AE | the adverse events rate and types of all enrolled patients, through study completion, an average of 1 year
  the adverse events of all enrolled patients

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China